CLINICAL TRIAL: NCT04822155
Title: The Social Gradient of Urban Noise Pollution and Its Effect on Pediatric and Adult Health
Status: Withdrawn | Type: Observational
Why Stopped: We did not have enough bandwidth to take on this project due to other project priorities.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 833334
Record Dates: First submitted 2021-03-04; First posted 2021-03-30 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Noise Exposure; Environmental Exposure; Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: Children between 11-17 years of age will be asked to participate in a home visit, where they respond to questions about certain actions or behaviors that affect their physical, emotional, or mental well-being (BRIEF-II and CBCL questionnaires). The child will also be asked to wear an actigraphy device on their wrist for 14 days while he/she sleeps to track their sleep quality.
- Adults: Adults, 18 years and older will be asked to participate in a home visit, where they respond to questions about certain actions or behaviors that affect your physical, emotional, or mental well-being (BRIEF-A and ABCL questionnaires). The adult will also be asked to wear an actigraphy device on their wrist for 14 days while he/she sleeps to track their sleep quality. Additionally, the adult will need to take their blood pressure 3 times per day for 14 days and record measurements.

SUMMARY:
The investigators pilot test an intervention to understand the spatial-temporal distribution of aggregated environmental noise exposure in Philadelphia and its impact on health.

DETAILED DESCRIPTION:
Noise pollution - sound created by human activities considered harmful to health - represents an oft- cited public concern, yet has taken a back seat to other environmental hazards. A limited number of observational studies demonstrate that chronic environmental noise exposure is associated with poor outcomes in adults and children, including cardiovascular disease, poor mental health, impaired sleep, and reduced cognitive performance in children. Further investigation and direct measurement at a community-level is needed to not only better understand the spatial-temporal distribution of aggregated environmental noise exposure and its impact on health, but also to lay the groundwork to develop and evaluate needed noise-reducing interventions.

The broad objective of this pilot proposal is to examine the social gradient of noise at a micro-spatial level in Philadelphia and evaluate its impact on the health of pediatric and adult local residents. Our multi-disciplinary team uniquely combines emerging digital and remote-sensing technologies, and expertise in place- based interventions to achieve the following specific aims: (AIM 1) Document the spatial-temporal distribution of environmental noise exposure across 24 Philadelphia neighborhoods with low, medium, and high socioeconomic status (SES), and (AIM 2) Explore the feasibility of evaluating the relationship between noise exposure and biometric health data - including sleep quality, cardiovascular metrics, and neurobehavioral profiles in pediatric and adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Residents living within 0.25 miles of the location of an external sound device
* Adults 18 years and older
* Children between 11-17 years of age
* Able to understand and respond to an oral interview in English

Exclusion Criteria:

* Unwilling to wear an Actigraphy device
* Adults unwilling to take blood pressure

Min Age: 11 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Our population includes adult (18 years and older) and adolescent (11-17 years) subjects living in target Philadelphia neighborhoods determined by noise profiles (AIM 1).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Environmental noise measurement of 24 Philadelphia neighborhoods using outdoor remote monitoring via International Electrotechnical Commission (IEC) | 30 days
  Environmental noise will be directly measured using outdoor remote monitoring via International Electrotechnical Commission (IEC) Class I portable sound level meter systems, which will allow for collection of comprehensive measurements (i.e. every second) over space and time. Noise will be measured for 30 days each at 24 sites, 8 each in low, medium, and high socioeconomic neighborhoods.
Measures of feasibility | 14 days
  Feasibility will be measured by the amount of usable remote biometric data collected.
Measures of acceptability | 14 days
  To measure acceptability, qualitative interviews will be conducted to provide insight on participants' experience with Actigraphy devices and sound devices in the home.

SECONDARY OUTCOMES:
Sleep duration using an Actigraphy device (adults and pediatric) | 14 days
  Sleep duration will be measured using an Actigraphy device, which helps assess sleep/wake patterns. The Actigraphy is a small, limb-worn activity monitor, typically placed on the wrist or ankle, designed for documenting physical movement associated with applications in psychological monitoring. The device is intended to monitor limb activity associated with movement during sleep.
Sleep quality using an Actigraphy device (adults and pediatric) | 14 days
  Sleep quality will be measured using an Actigraphy device, which helps assess sleep/wake patterns. The Actigraphy is a small, limb-worn activity monitor, typically placed on the wrist or ankle, designed for documenting physical movement associated with applications in psychological monitoring. The device is intended to monitor limb activity associated with movement during sleep.
Cardiovascular health (adults only) | 14 days
  This will be measured using ambulatory blood pressure monitoring three times per day.
Neurobehavioral measures (pediatric): BRIEF-II | 14 days
  This will be measured using the Behavior Rating Inventory of Executive Functions (BRIEF-II). The BRIEF-II evaluates children and adolescents with developmental and acquired neurological conditions. It consists of 63 questions on a Likert-type format with 0 ("Never"), 1 ("Sometimes"), 2 ("Often") that reflect the frequency to which the child being evaluated performs an indicated behavior. Higher scores indicate greater impairment in executive functioning.
Neurobehavioral measures (pediatric): CBCL | 14 days
  The Child Behavioral Checklist (CBCL) is a checklist parents complete to detect emotional and behavioral problems in children and adolescents. It consists of 113 questions, scored on a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often). The time frame for item responses is the past six months. The CBCL is computer scored, in which a trained professional needs to interpret the results.
Neurobehavioral measures (adults): BRIEF-A | 14 days
  This will be measured using the Behavior Rating Inventory of Executive Functions- Adult Version (BRIEF-A). The BRIEF-A captures views of an adult's executive functions or self-regulation in his or her everyday environment. It includes 75 items within nine nonoverlapping scales: Inhibit, Self-Monitor, Plan/Organize, Shift, Initiate, Task Monitor, Emotional Control, Working Memory, and Organization of Materials. All 75 items are rated in terms of frequency on a 3-point scale: 0 ("Never"), 1 ("Sometimes"), 2 ("Often"). Higher scores indicate greater impairment in executive functioning.
Neurobehavioral measures (adults): ABCL | 14 days
  The Adult Behavioral Checklist (ABCL) obtains information regarding an adult's adaptive functioning, problems and substance abuse. It consists of 132 questions on eight empirically based scales: Anxiety/Depression, Withdrawal, Somatic Complaints, Thought Problems, Attention Problems, Aggressive Behaviour, Rule Breaking Behaviour, Obsession-Compulsion. Responses are collected using three levels: "not true", "sometime true" and "often true".